CLINICAL TRIAL: NCT05212363
Title: Lower Leg Compression vs. a Walking Break on Blood Flow in Extended Video Game Play: A Pilot Study
Brief Title: Lower Leg Compression in Extended Video Game Play: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to financial cost.
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BHS-1664
Record Dates: First submitted 2021-09-01; First posted 2022-01-28 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Compression; Vein; Compression; Artery; Sedentary Behavior; DVT of Legs
Keywords: Esport; Gaming; Video games
MeSH Terms: conditions — Sedentary Behavior; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Twelve healthy collegiate esport players will be recruited for this single-arm pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Calf Compression (Experimental): Subjects will wear calf compression garments while video gaming for 2 hours. All subjects will undergo blood flow assessments before and after wearing lower leg graduated compression gear during their gaming session (i.e. compression during uninterrupted sitting).
  Interventions: Device: Lower extremity compression garments
- 6- minute Walk (Experimental): Subjects will game for 2 hours sitting and take a 6 minute walking break at the one hour period before resuming game play. All subjects will undergo blood flow assessments before and after taking an active break (i.e. 6-minute walk) during their gaming session.
  Interventions: Behavioral: Active break
- Continuous video game play (No Intervention): Subjects will game for 2 hours sitting with no break. All subjects will undergo blood flow assessments without wearing lower leg graduated compression gear or taking an active break during their gaming session (i.e. during uninterrupted sitting).

INTERVENTIONS:
Device: Lower extremity compression garments — Compression garments are used to exert external pressure on the lower extremities to reduce vascular wall tension and prevent gravity form pooling blood in the lower extremities which will improve venous return and lymphatic output. Following the resting measurements, subjects will be instructed to wear the garments and moved to the seated gaming position for 2 hours.
  Arms: Calf Compression
Behavioral: Active break — An active break is currently considered "gold standard" for increasing blood flow after prolonged sitting. The 6-minute walk will be conducted indoors next to the esport lab in the Wisser library at NYIT, Old Westbury. Participants will be asked to walk for 6 minutes on a flat surface back and forth following one hour of game play.
  Arms: 6- minute Walk

SUMMARY:
Compression garments are used to exert external pressure on the lower extremities to reduce vascular wall tension and prevent gravity form pooling blood in the lower extremities which will improve venous return and lymphatic output. Given the nature of video game play, sitting for prolonged periods of time without an active break is the perfect scenario to put these players at risk for deep vein thromboses (DVTs). Graduated compression wear may offer significant health benefits to this rapidly expanding sport. This study is essential to the formation of effective performance wear to reduce health risks in a gaming population.

DETAILED DESCRIPTION:
The use of compression wear has expanded from clinical use into the sports market. The recommendations to wear compression gear in athletes is based on improvement in venous blood flow which improves exchange of fresh blood and blood waste. The findings of research on its use to improve running performance has been mixed. Anecdotally, in 2001 Allen Iverson of the National Basketball Association (NBA) wore a compression arm sleeve to prevent swelling and provide relief of bursitis in his elbow. Lebron James of the NBA and London marathon runner Paul Radcliffe both swear by compression gear. In the 2016 Olympics, it was estimated that 90% of athletes used some form of compression performance gear. (1) The compression wear sports industry market is a billion-dollar industry projected to be worth 3.96 billion dollars by 2022.(1) Clinicians traditionally prescribe compression gear to reduce the incidence of deep vein thrombosis (DVT). Deep vein thrombosis (DVT) is a blood clot that forms in a vein. Usually this clot forms in the leg or pelvic veins. Symptoms of DVT's can vary from swelling in a particular region, sensitivity, and on some occasions, there may not be any clinical signs. in hospital patients who are immobile or undergo surgery and that are at increased risk for DVT's. Compression gear also reduces the risk of DVT's in a variety of other health and environmental conditions which include, but not limited to, long periods of being immobile, older age, illness and prolonged sitting.(2) These clots can become life threatening as they can travel to the lungs, potentially leading to a pulmonary embolism (PE) and death. (2,3) Dr. Beasley coined the term "e-thrombosis" hypothesizing that the increase in computer use for work and decreased physical activity would lead to an increase in DVT's and PE's brought on by immobility and prolonged sit time.(4) Fast forward to the present where esports and video game use has exploded at an astronomical rate, and Dr. Beasley's theory would be fortified by many case studies and clinical studies documenting computer use is a major contributor to DVT. There have been over 22 documented cases of DVT's brought on by excessive gaming in the past few years. (5) Although DVT's are not the norm, gamers have nearly double the risk of developing a thrombolytic event as compared to non-gamers.(6) A triad of physiological changes has been proposed that increase the risk of DVT. The first one is changes in blood flow, the second is changes in the blood itself, and lastly is the integrity of the endothelial lining of the blood vessels. Typically, when we are moving, skeletal muscle goes through contraction and relaxation to help pump blood throughout the body and against gravity. When in a sitting position the velocity of blood flow in the upwards direction (against gravity) is reduced. After 3 hours of uninterrupted prolonged sitting, femoral artery blood flow can decline up to 50%. (7,8) Even in children 7-10 years of age, femoral artery blood flow decreased by 33%.(9) This decreased blood flow disturbs homeostasis, can result in blood pooling in the lower extremities, creates procoagulant changes in the blood, endothelial activation and is the primary cause of DVT. Several studies have demonstrated that a 3 minute light walking break at 30 minutes can increase popliteal blood flow by up to 30% and improve cerebral blood flow.(10-12) In a recent study by the current author (DiFrancisco-Donoghue et al.), it was reported that the average collegiate gamer sits 4-8 hours daily while practicing their craft.(13) These extended hours of sitting and play time can vary extensively among recreational gamers as reported in table 1 by Lippi et al.(5) Based on these findings, the authors' current study observed a 6 minute walking break compared to a 6-minute resting break in prolonged gamers on cognitive function. This study was conducted virtually during the pandemic and currently under review. The 6-minute break was based on findings by Chrismas et al. who found a 3-minute walking break at 30 minutes improved attention and executive function.(12) Breaking up an esport game every 30 minutes is not reasonable, therefore we chose to break at 60 minutes of play using the cumulative time of 6 minutes. This study demonstrated an improvement in executive function in the 6-minute walking break compared to the resting break following prolonged game play. Due to the pandemic, since the investigators were unable to collect physiological data on participants, we are adapting the same protocol without testing executive function, but rather observing the physiological changes that occur from a walking break and from using compression wear.

Athletes in various sports wear compression garments with the assumption that it will improve performance and facilitate muscle recovery. Most modern compression gear is marketed toward athletes use 'graduated compression'. This means that the highest amount of pressure is on the most distal parts of your body (e.g ankles if you are using lower body compression) and the pressure gradually reduces as it moves up toward your body. Compression wear varies in pressure range. The measurement is measured in mmHg and light compression can range from 18-21 mmHg, moderate 23-32 mmHg, strong 34-46 mmHg and > 49 mmHg very strong. (14) Most over the counter athletic compression garments range from 18-21 mmHg.

Twelve healthy collegiate esport players will be recruited for this pilot study. This study will be a randomized cross-over design trial which will require subjects to come to the NYIT esport gaming lab at least one hour post prandial for 3 testing days lasting 2.5 hours. The room will be kept temperature controlled for each subject and kept within 2-3 degrees Celsius each testing day. Subjects will sign a written consent and then rest quietly sitting in the gaming chair for 10 minutes. After the rest period, popliteal artery blood flow velocity, flow-mediated dilation (FMD) and shear rate will be assessed at rest using a doppler ultrasound bilaterally. Carotid artery blood flow will also be measured. Blood pressure and heart rate will be assessed.

Testing day 1: Following the 10 minute rest/measurement phase, all subjects will play continuous for 2 hours on day one with no break. During the seated period measurements will be taken bilaterally at 30 minutes, 1 hour and 2 hours on the legs and the carotid artery. The popliteal artery is located behind the knee. The subjects will extend the leg slightly to allow the technician to take the measurements while remaining seated. The carotid artery is located laterally on the neck region. In the current study, the measurements will be conducted while seated by the radiology technician.

Testing day 2: This study will use lower leg graduated compression garments with a compression between 20-30 mmHg. Each leg will be fitted according to manufacturer instructions. Following the resting measurements, subjects will be instructed to wear the garments and moved to the seated gaming position for 2 hours. During the seated period blood flow velocity, FMD and shear rate will be taken within the first 10 minutes upon sitting as well as 30 minutes, 1 hour and 2 hours on both compression legs and the carotid artery.

Testing day 3: The 6-minute walk will be conducted indoors next to the esport lab in the Wisser library at NYIT, Old Westbury. Participants will be asked to walk for 6 minutes on a flat surface back and forth following one hour of game play. All blood flow measures will be taken prior to the subject standing and conducting the walk. An investigator will be timing them. Prior to the walk the participants will be shown the 6-20 BORG Rating of Perceived Exertion Scale (RPE) that will be held up by the investigators. This RPE is a validated scale to measure how hard a person feels they are working during physical activity and has been validated to correlate heart rate and perceived effort during active videogame play.(15) The subjects' heart rate will also be taken by brachial pulse prior to walking and following the 6-minute walk. Upon return to the gaming lab, all blood flow measurements will be repeated. The subjects will then play for another hour where all measurements will be repeated following the gaming session. Upon completion of testing on day 3, subjects will be given a short survey regarding their perceptions of wearing the compression garments.

ELIGIBILITY:
Inclusion Criteria:

1. Ranked esport player with over 500 hours in their game.
2. Non-smoker.
3. No history of heart disease, pulmonary disease, or metabolic disease including diabetes.
4. Taking any prescribed or over the counter medications that would influence metabolic outcomes or blood viscosity.

Exclusion Criteria:

1. Peripheral neuropathy or any other condition that impacts skin sensation.
2. A history of a peripheral arterial bypass grafting.
3. Peripheral artery disease.
4. Skin infection.
5. Dermatitis with oozing or fragile skin.
6. Current leg swelling
7. Pulmonary edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Popliteal artery blood flow velocity | 2 hours
  A B0MJ18Philips L9-3 Transducer will be used to measure popliteal artery blood velocity at rest, and every 30 minutes for 120 minutes during prolonged gaming
Popliteal artery blood Volume | 2 hours
  A B0MJ18Philips L9-3 Transducer will be used to measure popliteal artery blood volume at rest, and every 30 minutes for 120 minutes during prolonged gaming
Popliteal artery Transverse Diameter | 2 hours
  A B0MJ18Philips L9-3 Transducer will be used to measure popliteal artery transverse diameter at rest, and every 30 minutes for 120 minutes during prolonged gaming

SECONDARY OUTCOMES:
Compression garment and Esport performance perception survey | 2 hours
  Subjects will be given a likert scale on their perception of wearing compression garments while gaming following completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donoghue, Principal Investigator — Director of Clinical Research
Locations (1):
- New York Institute of Technology College of Osteopathic Medicine, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Book J, Prince CN, Villar R, Hughson RL, Peterson SD. Investigating the impact of passive external lower limb compression on central and peripheral hemodynamics during exercise. Eur J Appl Physiol. 2016 Apr;116(4):717-27. doi: 10.1007/s00421-016-3331-0. Epub 2016 Jan 25. PMID 26811062
- [Background] Beasley R, Raymond N, Hill S, Nowitz M, Hughes R. eThrombosis: the 21st century variant of venous thromboembolism associated with immobility. Eur Respir J. 2003 Feb;21(2):374-6. doi: 10.1183/09031936.03.00039403. PMID 12608454
- [Background] Lippi G, Mattiuzzi C, Favaloro EJ. e-thrombosis: epidemiology, physiopathology and rationale for preventing computer-related thrombosis. Ann Transl Med. 2018 Sep;6(17):344. doi: 10.21037/atm.2018.09.03. PMID 30306083
- [Background] Pearce L. Playing with danger. Nurs Stand. 2012 Aug 29-Sep 4;26(52):25. doi: 10.7748/ns.26.52.25.s24. PMID 23061127
- [Background] Restaino RM, Holwerda SW, Credeur DP, Fadel PJ, Padilla J. Impact of prolonged sitting on lower and upper limb micro- and macrovascular dilator function. Exp Physiol. 2015 Jul 1;100(7):829-38. doi: 10.1113/EP085238. Epub 2015 Jun 10. PMID 25929229
- [Background] McManus AM, Ainslie PN, Green DJ, Simair RG, Smith K, Lewis N. Impact of prolonged sitting on vascular function in young girls. Exp Physiol. 2015 Nov;100(11):1379-87. doi: 10.1113/EP085355. Epub 2015 Oct 7. PMID 26370881
- [Background] Wennberg P, Boraxbekk CJ, Wheeler M, Howard B, Dempsey PC, Lambert G, Eikelis N, Larsen R, Sethi P, Occleston J, Hernestal-Boman J, Ellis KA, Owen N, Dunstan DW. Acute effects of breaking up prolonged sitting on fatigue and cognition: a pilot study. BMJ Open. 2016 Feb 26;6(2):e009630. doi: 10.1136/bmjopen-2015-009630. PMID 26920441
- [Background] Carter SE, Draijer R, Holder SM, Brown L, Thijssen DHJ, Hopkins ND. Regular walking breaks prevent the decline in cerebral blood flow associated with prolonged sitting. J Appl Physiol (1985). 2018 Sep 1;125(3):790-798. doi: 10.1152/japplphysiol.00310.2018. Epub 2018 Jun 7. PMID 29878870
- [Background] Chrismas BCR, Taylor L, Cherif A, Sayegh S, Bailey DP. Breaking up prolonged sitting with moderate-intensity walking improves attention and executive function in Qatari females. PLoS One. 2019 Jul 12;14(7):e0219565. doi: 10.1371/journal.pone.0219565. eCollection 2019. PMID 31299061
- [Background] DiFrancisco-Donoghue J, Balentine J, Schmidt G, Zwibel H. Managing the health of the eSport athlete: an integrated health management model. BMJ Open Sport Exerc Med. 2019 Jan 10;5(1):e000467. doi: 10.1136/bmjsem-2018-000467. eCollection 2019. PMID 30792883
- [Background] Berszakiewicz A, Sieron A, Krasinski Z, Cholewka A, Stanek A. Compression therapy in venous diseases: physical assumptions and clinical effects. Postepy Dermatol Alergol. 2020 Dec;37(6):842-847. doi: 10.5114/ada.2019.86990. Epub 2019 Jul 26. PMID 33603600
- [Background] Pollock BS, Barkley JE, Potenzini N, Desalvo RM, Buser SL, Otterstetter R, Juvancic-Heltzel JA. Validity of Borg Ratings of Perceived Exertion During Active Video Game Play. Int J Exerc Sci. 2013 Apr 15;6(2):164-170. doi: 10.70252/XGRF9788. eCollection 2013. PMID 27293499
- [Background] Restaino RM, Walsh LK, Morishima T, Vranish JR, Martinez-Lemus LA, Fadel PJ, Padilla J. Endothelial dysfunction following prolonged sitting is mediated by a reduction in shear stress. Am J Physiol Heart Circ Physiol. 2016 Mar 1;310(5):H648-53. doi: 10.1152/ajpheart.00943.2015. Epub 2016 Jan 8. PMID 26747508
- See also: Compression Therapy Market Size, Growth, Trends | Global Report 2026 [Internet]. [cited 2021 Apr 23]. — https://www.fortunebusinessinsights.com/compression-therapy-market-102689